CLINICAL TRIAL: NCT02070471
Title: A Multicenter, Randomized, Parallel Group, Double-Blind, Placebo-Controlled Phase 2 Study to Evaluate the Efficacy, Safety and Pharmacokinetics of Intravenous Single Injection LC28-0126 Immediately Before PCI (Percutaneous Coronary Intervention) in Patients With STEMI(ST-segment Elevation Myocardial Infarction)
Brief Title: Phase 2 Study to Evaluate the Efficacy, Safety and PK of Intravenous Single Injection LC28-0126 Immediately Before PCI in STEMI Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: LG Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LG-CYCL002
Record Dates: First submitted 2014-02-21; First posted 2014-02-25 (Estimated); Last update posted 2016-05-10 (Estimated); Status verified 2015-09

CONDITIONS: ST-segment Elevation Myocardial Infarction
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- LC28-0126 Dose A (Experimental): LC28-0126 Dose A
  Interventions: Drug: LC28-0126 Dose A
- LC28-0126 Dose B (Experimental): LC28-0126 Dose B
  Interventions: Drug: LC28-0126 Dose B
- LC28-0126 Dose C (Experimental): LC28-0126 Dose C
  Interventions: Drug: LC28-0126 Dose C
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Placebo
  Arms: Placebo
Drug: LC28-0126 Dose A — LC28-0126 Dose A
  Arms: LC28-0126 Dose A
Drug: LC28-0126 Dose B — LC28-0126 Dose B
  Arms: LC28-0126 Dose B
Drug: LC28-0126 Dose C — LC28-0126 Dose C
  Arms: LC28-0126 Dose C

SUMMARY:
Evaluate the efficacy, Safety and Pharmacokinetics of Intravenous single injection LC28-0126 immediately before PCI (Percutaneous Coronary Intervention) in Patients with STEMI (ST-segment Elevation Myocardial Infarction)

ELIGIBILITY:
Inclusion Criteria:

* Age between 20 and 75
* Within 12 hours after the onset of chest pain
* ST-segment elevation of more than 0.1 mV in two contiguous leads or new LBBB(left bundle-branch block) patients
* Signed for written informed consent

Exclusion Criteria:

* Left Main disease
* Multi-vessel disease

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-01; Primary Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
AUC of CK-MB for 72 hours post PCI | pre PCI, PCI 0h, 6h, 12h, 18h, 24h, 48h, 72h

SECONDARY OUTCOMES:
AUC of Troponin I and CK for 72h post PCI | pre PCI, PCI 0h, 6h, 12h, 18h, 24h, 48h, 72h
Infarct size and myocardial function assessed by CMR and Echocardiogram | Day 4, 30

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea